CLINICAL TRIAL: NCT04626817
Title: Effect of Oral Isotretinoin on Muscle Strength in Patients With Acne Vulgaris: A Prospective Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cevriye Mülkoğlu (Other)
Responsible Party: Sponsor-Investigator, Cevriye Mülkoğlu, Medical Doctor in Department of Physical Medicine and Rehabilitation, Ankara Training and Research Hospital
Organization: Ankara Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Ankara TRH
Record Dates: First submitted 2020-11-03; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Muscle Strength
Keywords: Isotretinoin; muscle strength; isokinetic; creatinine phosphokinase

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isotretinoin receiving group (Active Comparator): Isotretinoin receiving group for acne vulgaris
  Interventions: Device: Isokinetic device (Biodex System 4)
- Local treatment receiving group (Placebo Comparator): Local treatment receiving group for acne vulgaris
  Interventions: Device: Isokinetic device (Biodex System 4)

INTERVENTIONS:
Device: Isokinetic device (Biodex System 4) — The measurement of muscle strength with isokinetic device
  Other Names: serum creatinine phosphokinase level

SUMMARY:
BACKGROUND: Musculoskeletal side effects related to isotretinoin are frequently reported. This study aimed to investigate the effect of oral isotretinoin treatment on muscle strength. Our second aim was to evaluate whether there was a correlation between the serum creatine phosphokinase (CPK) level, a specific marker of muscle breakdown, and muscle strength.

METHODS: This study included 30 patients who presented to our hospital and were started on oral isotretinoin treatment for acne vulgaris and 30 patients in the control group who were given local treatment. Age, gender, height and weight of the patients were recorded, and the body mass index (BMI) was calculated. The hamstring and quadriceps muscle strengths of the non-dominant side were evaluated in all patients using an isokinetic dynamometer, and the peak torque (PT) values were recorded. In the isotretinoin group, isokinetic measurements were performed again in those that completed six-month drug treatment and compared with the initial PT values.

DETAILED DESCRIPTION:
BACKGROUND: Musculoskeletal side effects related to isotretinoin are frequently reported. This study aimed to investigate the effect of oral isotretinoin treatment on muscle strength. Our second aim was to evaluate whether there was a correlation between the serum creatine phosphokinase (CPK) level, a specific marker of muscle breakdown, and muscle strength.

METHODS: This study included 30 patients who presented to our hospital and were started on oral isotretinoin treatment for acne vulgaris and 30 patients in the control group who were given local treatment. Age, gender, height and weight of the patients were recorded, and the body mass index (BMI) was calculated. The hamstring and quadriceps muscle strengths of the non-dominant side were evaluated in all patients using an isokinetic dynamometer, and the peak torque (PT) values were recorded. In the isotretinoin group, isokinetic measurements were performed again in those that completed six-month drug treatment and compared with the initial PT values.

ELIGIBILITY:
Inclusion Criteria:

* being aged 18-45 years
* receiving isotretinoin treatment for the isotretinoin group
* not having used isotretinoin within the last year for the control group

Exclusion Criteria:

* chronic kidney or liver disease,
* uncontrolled hypertension, heart failure,
* malignancy,
* thyroid and bone diseases (e.g., hyperparathyroidism and osteomalacia),
* use of drugs that may affect skeletal metabolism (e.g., corticosteroids, heparin, and anticonvulsants),
* a history of trauma and/or surgery in the lower extremities.
* Patients who discontinued or terminated their isotretinoin treatment were not included in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
The hamstring and quadriceps muscle strengths of the non-dominant lower extremity | 6 months
  peak torque values
creatinine phosphokinase | 6 months
  serum creatinine phosphokinase level

CONTACTS AND LOCATIONS:
Overall Officials: Cevriye Mülkoglu, Principal Investigator — Saglik Bakanligi Ankara Egitim ve Arastirma Hastanesi
Locations (1):
- Ankara Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Mulkoglu C, Karaosmanoglu N. Effect of oral isotretinoin on muscle strength in patients with acne vulgaris: a prospective controlled study. BMC Pharmacol Toxicol. 2021 Mar 20;22(1):17. doi: 10.1186/s40360-021-00483-0. PMID 33743831